CLINICAL TRIAL: NCT07282873
Title: A Phase I/II, Open-label, Multicenter Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of the TEAD Inhibitor TYK-01054 Capsules in Patients With Locally Advanced or Metastatic Advanced Solid Tumors
Brief Title: Study of TYK-01054 Capsules in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TYK Medicines, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TYKM1408101
Record Dates: First submitted 2025-11-18; First posted 2025-12-15 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumor Malignancies; Malignant Mesothelioma (MM)
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TKY-01054 (Experimental): TKY-01054，orally administered daily
  Interventions: Drug: TYK-01054

INTERVENTIONS:
Drug: TYK-01054 — TKY-01054 will be administered orally at a starting dose of 25 mg in 21-day cycles. If well tolerated, dose expansion will proceed in the recommended dose for expansion (RDE) and RDE-1 until the recommended Phase II dose (RP2D) is determined.

SUMMARY:
This study is to evaluate the safety, tolerability, pharmacokinetics, and antitumor activity of the TEAD inhibitor TYK-01054 capsules in patients with locally advanced or metastatic advanced solid tumors

DETAILED DESCRIPTION:
Dose Escalation (Part A) will employ an accelerated titration design combined with a "3 + 3" design to evaluate the safety and pharmacokinetic (PK) profile of TYK-01054 in patients with mesothelioma and/or metastatic solid tumors who are resistant to standard therapy or for which no effective standard therapy is available. Dose escalation phase comprises a single-dose stage (7 days) and a continuous dosing stage. Accelerated titration will switch to the conventional 3+3 design as soon as any patient experiences a ≥Grade 2 TYK-01054-related toxicity or when the second patient at any dose level completes the first cycle without dose-limiting toxicity (DLT). Dose escalation will continue until the Maximum Tolerated Dose (MTD), Recommended Dose for Expansion (RDE), or a suitable intermittent dosing regimen is determined. The RDE(s) selected in Part A will be carried forward into the dose optimisation phase.

Dose Optimization (Part B) will further assess safety and PK, and will evaluate preliminary anti-tumor activity at two RDE levels. Approximately 40 patients with four target indications will be enrolled and randomised 1:1 to receive either RDE or RDE-1. Based on PK, safety, and all cumulative data, the Study Review Committee (SRC) will determine the dose for the Part c (i.e., the Recommended Phase 2 Dose, RP2D).

Cohort Expansion (Part C) includes four cohorts.

* Cohort 1: Advanced (unresectable or metastatic) malignant mesothelioma(MM); regardless of NF2 mutation status or other Hippo pathway abnormalities.
* Cohort 2: Advanced (unresectable or metastatic) Small-cell lung cancer (SCLC) that has progressed after first-line therapy.
* Cohort 3: Advanced (unresectable or metastatic) Head-and-neck squamous-cell carcinoma (HNSCC) that has progressed after first-line systemic therapy.
* Cohort 4: Advanced (unresectable or metastatic) solid tumours; priority will be given to colorectal cancer (CRC), pancreatic ductal adenocarcinoma (PDAC), non-small-cell lung cancer (NSCLC), and epithelioid haemangioendothelioma (EHE).

Cohorts 2-4 require that patients also have abnormalities in the Hippo signaling pathway, NF2, MST1/2, LATS1/2, FAT1 mutations/alterations or YAP/TAZ fusion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 years old
2. Histologically or cytologically confirmed incurable, locally advanced or metastatic advanced solid tumors. All participants are required to provide results of Hippo signaling pathway gene testing; however, this requirement is not a mandatory inclusion criterion for Dose Escalation (Part A) and EHE patients.
3. Advanced solid tumors must have progressed after receiving at least one standard first-line anti-tumor therapy, OR demonstrate intolerance to standard therapy, OR Lack of standard treatment.
4. Patients should have at least 1 measurable lesion as per RECIST v1.1 or mRECIST v1.1.
5. Adequate organ function, including hepatic, renal, cardiovascular, astrointestinal,respiratory, and hematopoietic systems.
6. ECOG 0-1，
7. Life expectancy of >3 months.
8. Willing and able to comply with all aspects of the protocol.

Exclusion Criteria:

1. History of other malignancy, except for:

   Non-melanoma skin cancer (basal cell carcinoma or squamous cell carcinoma) that is non-invasive and has been effectively controlled with no recurrence or metastasis for 5 years, Papillary thyroid carcinoma, Carcinoma in situ of the cervix, Ductal carcinoma in situ of the breast.
2. Unstable brain metastases,such as:

   Patients requiring urgent neurosurgical intervention for CNS complications, Presence of symptomatic spinal cord compression due to tumor, Presence of leptomeningeal disease (carcinomatous meningitis).
3. Presence of pleural effusion, pericardial effusion, or ascites that, in the investigator's judgment, cannot be stably controlled by repeated drainage or other methods.
4. Clinically significant renal disease.
5. Clinically significant cardiovascular disease, including but not limited to myocardial infarction, unstable angina, congestive heart failure (NYHA Class ≥ II), or uncontrolled arrhythmias.
6. Patients with uncontrolled infectious diseases, such as immunodeficiency disorders (e.g., HIV) or active hepatitis B or C infection; chronic hepatitis B or C carriers without symptoms are excluded from this criterion.
7. Known or suspected hypersensitivity to TYK-01054 or any of its excipients, or to compounds of similar chemical class.
8. Patients who have previously received a TEAD inhibitor.
9. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | Up to approximately 28 days
  Numbers of participants experiencing AEs which are defined as DLTs classfied by CTCAE v6.0
Maximum tolerated dose（MTD） | Through the Dose Escalation phase, approximately 12 months
  The maximum dose when DLT% ≤ 33% during the DLT observation period
Number of participants who experience one or more adverse events (AEs) | From Baseline up to 28 days after the end of the treatment
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Recommended Dose for Expansion(RDE) | Through the Dose Escalation Phase, approximately 24 months
  Recommended Dose for Expansion
Recommended Phase 2 Dose（RP2D） | Within 28 days of the last patient dosed in the Dose Optimization stage
  The RP2D is defined as the dose level chosen for the dose expansion arms, based on safety, tolerability, efficacy, pharmacokinetics (PK), and pharmacodynamic (PD) data collected during the dose escalation portion of the study.

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of TYK-01054 | Through the Dose Escalation stage and Dose Optimization stage, approximately 24 month
  Based on the plasma concentration ofTYK-01054
Evaluate the effectiveness of TYK-01054 | Approximately 36 months
  Efficacy evaluation will be determined by RECIST v1.1 or modified RECIST v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No